CLINICAL TRIAL: NCT07168824
Title: An Open Label Trial Evaluating the Efficacy of Lacticaseibacillus Paracasei PS23 on Cognition
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chi-Chang Huang (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chi-Chang Huang, Dean of Research and Development, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-25-061-A2
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Subjective Cognitive Decline (SCD)
Keywords: Subjective Cognitive Decline; Mild cognitive impairment; probiotics; dietary supplement
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotics (Experimental): Lacticaseibacillus paracasei PS23 one capsule daily for 12 weeks
  Interventions: Dietary Supplement: Lacticaseibacillus paracasei

INTERVENTIONS:
Dietary Supplement: Lacticaseibacillus paracasei — one capsule daily for 12 weeks
  Other Names: PS23

SUMMARY:
This open label study aims to evaluate whether the consumption of probiotics can improve symptoms and overall quality of life in individuals experiencing cognitive decline symptoms, as well as to evaluate the effects of probiotics on blood-related biomarkers.

DETAILED DESCRIPTION:
Lacticaseibacillus paracasei PS23 (PS23) is a specific strain of probiotic bacteria known for its potential health benefits, particularly in the context of aging and muscle health. Research suggests that it may improve cognitive function, reduce age-related muscle loss, and modulate the gut microbiota. Probiotic supplements like PS23 are being explored as potential therapeutic agents for age-related cognitive deficits. A prior study showed that PS23 supplementation delayed age-related cognitive decline in mice. Additionally, PS23 has shown antidepressant-like effects and has been found to enhance physical performance and promote muscle recovery following injury.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 to 85 years who self-report experiencing signs of cognitive decline.
* No prior diagnosis of dementia or Alzheimer's disease (AD).
* Willing and able to comply with study assessments and requirements, and provide written informed consent.

Exclusion Criteria:

* Use of antibiotics or probiotic powder, capsules, or tablets within the past month.
* Currently undergoing antibiotic treatment.
* Known allergy to dairy products.
* Presence of immunodeficiency or impaired immune function.
* Diagnosis of small intestinal bacterial overgrowth (SIBO).
* Determined unsuitable by the investigator, for example, initiation of any new medication or therapy during the study period, particularly those related to memory impairment or cognitive decline.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological measures Changes in CANTAB® in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  Cambridge Neuropsychological Test Automated Battery (CANTAB®) includes computerized tests that are correlated to neural networks and have demonstrated high sensitivity in detecting changes in neuropsychological performance.

SECONDARY OUTCOMES:
Changes in Chinese version of Trail Making Test (TMT) in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  The Trail Making Task (TMT) is a neuropsychological test consisting of two parts that assesses executive function, visual attention, speed of processing, and cognitive flexibility. In Part A, the participant connects 25 numbered circles in sequential numerical order (1 to 25) as quickly and accurately as possible. TMT-B with sequential numbers in the Chinese characters substituting for the English alphabetical sequence, replaced numbers and letters of the TMT-B by circles and squares with numbers, modified the TMT-B with the Chinese zodiacs substituting for the English alphabet
Changes in Chinese version of Stroop color words test(SCWT) in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  The Stroop Color Words test (SCWT) was used to evaluate the dominant inhibition in executive function
Changes in Geriatric Depression Scale in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  The Geriatric Depression Scale (GDS) is a screening tool for depression in older adults (55+), consisting of a short, yes/no questionnaire about feelings over the past week. Scores range between 0 and 30 points. Higher scores indicate more severe depressive symptoms.
Changes in Anxiety Disorder Assessment (GAD-7) in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  The Generalised Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day"
Changes in The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 (QLESQ-16) in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 is a valid, reliable self-report instrument for assessing quality of life. The minimum raw score on the Q-LES-Q-16 is 14, and the maximum score is 70, higher scores mean a better outcome.
Changes in Patient Global Impression scales of Improvement rated by patient （PGI-C) in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  The PGIC consists of one item taken from the clinical global impression and adapted to the patient. The minimum total score possible is 1 and the maximum total score possible is 7. Higher values represent a worse outcome.
Changes in pTau-217 in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  Recent, research studies have shown that plasma levels of p-Tau 217 are elevated in AD patients1,2. Additionally, it has been demonstrated that plasma p-Tau 217 levels are increased in the early stages of the AD continuum and are correlated with amyloid-PET positivity.
Changes in Plasma Aβ40 and Aβ42 in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  Plasma Aβ42/Aβ40 is sensitive to early cerebral amyloid accumulation and predicts risk of cognitive decline across the Alzheimer's disease spectrum
Changes in Brain-derived neurotrophic factor (BDNF) in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  Brain-derived neurotrophic factor (BDNF) plays an important role in neuronal survival and growth, serves as a neurotransmitter modulator, and participates in neuronal plasticity, which is essential for learning and memory.
Changes in Glial Fibrillary Acidic Protein (GFAP) in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  Glial fibrillary acidic protein (GFAP), an astrocytic cytoskeletal protein, can be measured in blood samples, and has been associated with Alzheimer's disease (AD).
Changes in Neurofilament Light (NfL) in 40 subjects after probiotic intervention | baseline to 12 weeks assessed
  Neurofilament light chain (NfL) is a structural protein that normally helps support the shape and function of brain cells. In Alzheimer's disease (AD), brain cells are damaged, which causes the brain to shrink (atrophy), and symptoms such as declining cognition to occur.
Changes in Mandarin Subjective Cognitive Decline Scale (SCDS) in 40 subjects after probiotic intervention | screening, baseline to 12 weeks assessed
  Self-reported questionnaire consisting of 14 items assessing perceived decline in memory, attention, language, planning, orientation, and other cognitive domains. Responses are typically rated on a Likert scale (e.g., 0 = "Never" to 4 = "Very frequently"), with total scores ranging from 0 to 56-higher scores indicate greater subjective cognitive complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Chang Huang, PhD, Principal Investigator — National Taiwan Sport University
Locations (1):
- Graduate Institute of Sports Science, National Taiwan Sport University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided